CLINICAL TRIAL: NCT06963242
Title: Accuracy of Dynamic Navigation System in Implant Surgery for Full Arch Prosthesis
Brief Title: Evaluating the Accuracy of Dynamic Navigation in Implant Surgery for Full Arch Prosthesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Tran Cao Nhiem, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24384-DHYD
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Accuracy of Dynamic Navigation System in Implant Placement for Full Arch Prosthesis Rehabilitation
Keywords: Dynamic Navigation; Implant placement surgery; Full arch prosthesis; Surgical guide; Implant rehabilitation; Fully edentulous; Computer-assisted surgery; Surgical navigation; Implant accuracy; Tooth-based landmark; Screw-based landmark

STUDY DESIGN:
Intervention Model Description: This is a parallel design study that compares two intervention groups. Group 1 uses bone screws (4-6 screws) as reference landmarks for dynamic navigation-guided implant placement, while Group 2 uses remaining teeth as reference landmarks. Both groups undergo the same surgical procedure, and the study evaluates the accuracy of implant placement with dynamic navigation. The interventions are carried out in parallel, and the results will be compared between the two groups to assess the effectiveness of each reference system in implant placement for full arch prosthesis rehabilitation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bone Screw Group (Group 1) (Experimental): In this arm, participants will undergo implant placement using a dynamic navigation system. Bone screws (4-6 screws) will be placed in the jaw arch as reference points to ensure accurate implant placement. The primary objectives are to measure the deviation in implant placement compared to the planned data and to assess the surgery time required for implant placement using this system. The results will be compared with those from Group 2, where landmarks are based on remaining teeth to be extracted, to evaluate the accuracy and time efficiency between the two approaches.
  Interventions: Device: Dynamic Navigation System for Implant Placement Using Bone Screws as Landmarks
- Tooth Landmark Group (Group 2) (Experimental): In this arm, participants will undergo implant placement using a dynamic navigation system. Landmarks based on remaining teeth to be extracted will be used as reference points to ensure accurate implant placement. The primary objectives are to measure the deviation in implant placement compared to the planned data and to assess the surgery time required for implant placement using this system. The results will be compared with those from Group 1, where bone screws were placed as landmarks, to evaluate the accuracy and time efficiency between the two approaches.
  Interventions: Device: Dynamic Navigation System for Implant Placement Using Remaining Teeth as Landmarks

INTERVENTIONS:
Device: Dynamic Navigation System for Implant Placement Using Bone Screws as Landmarks — This study uses a dynamic navigation system for implant placement in fully edentulous patients requiring full arch prosthesis rehabilitation. The system incorporates bone screws (placed as reference points on the jaw arch) to guide the accurate placement of implants. Unlike traditional freehand implant placement, this dynamic navigation system aims to minimize deviation from the planned implant positions while also reducing the time required for the surgical procedure. The results will be compared to a group where landmarks are based on remaining teeth to assess accuracy and time efficiency of the system.
  Arms: Bone Screw Group (Group 1)
Device: Dynamic Navigation System for Implant Placement Using Remaining Teeth as Landmarks — In this arm, participants will undergo implant placement using a dynamic navigation system, where the reference points for implant positioning are based on the remaining teeth to be extracted. This approach, in contrast to the bone screw method used in Group 1, relies on the teeth that will be removed as landmarks to guide the accuracy of implant placement. The primary goal is to evaluate the accuracy of the implant placement and the time required for the procedure using this method. The results from this group will be compared to those from Group 1, where bone screws are placed as reference points, to assess the accuracy and time efficiency of both approaches.
  Arms: Tooth Landmark Group (Group 2)

SUMMARY:
Study Objective:

This study aims to evaluate the accuracy of the Dynamic Navigation System in performing implant placement for full arch prosthesis rehabilitation. This system uses landmarks, including bone screws fixed to the bone (Group 1), and landmarks on remaining teeth to be extracted (Group 2), to accurately determine the placement of the implants

Participants:

Patients aged 18 and older, who have total tooth loss or partial tooth loss, and are candidates for full arch implant-supported prosthesis rehabilitation, are invited to participate, provided they meet the necessary health requirements for surgery.

Group 1: Patients who have total tooth loss or partial tooth loss but do not meet the following conditions:

1. Having at least 3 remaining teeth or roots with mobility no greater than grade 1, and
2. The remaining teeth are distributed with at least 1 tooth in the front and 1 tooth in the back on each side of the arch. These patients will have bone screws placed on the bone to serve as landmarks for implant placement using the dynamic navigation system.

Group 2: Patients who have at least 3 remaining teeth, all with mobility no greater than grade 1, and at least one tooth in the front and one in the back on each side of the arch. These teeth will serve as landmarks for implant placement.

Study Methodology:

Group 1: Patients who have total or partial tooth loss, and do not meet the conditions of having at least 3 remaining teeth with mobility no greater than grade 1, and having at least one tooth in the front and one in the back on each side, will have bone screws placed on the bone as landmarks for implant placement.

Group 2: Patients with at least 3 remaining teeth with mobility no greater than grade 1, and at least one tooth in the front and one in the back on each side, will use these teeth as landmarks for implant placement.

After surgery, the implant deviation from the planned implant data will be evaluated to assess the accuracy of implant placement.

Factors such as implant position deviation, surgery time, and complications will be evaluated to compare the effectiveness between the two groups.

Benefits and Risks:

1. Benefits:

   1. Improved accuracy in implant placement using the Dynamic Navigation System.
   2. Cost of using the Dynamic Navigation System and the cost of bone screws for patients without sufficient remaining teeth are covered by the study.
   3. Scientific contribution to improving implant placement methods for future patients.
2. Risks:

   1. Surgical risks including infection, pain, swelling, and potential implant failure, which can occur even without the use of the dynamic navigation system.
   2. Radiation exposure from imaging tests, particularly CBCT scans, will be required. The radiation exposure is minimal and within safe limits.
   3. Slight increase in surgery time, typically 2-5 minutes longer than traditional surgery, for preparation and calibration of the navigation system to ensure its proper functionality.
   4. For Group 1 participants, bone screws (4-6 screws) will be placed along the jaw arch where the implants are to be positioned.

DETAILED DESCRIPTION:
Study Overview:

Full arch implant surgery is a highly effective treatment for patients with total or partial tooth loss. However, determining the precise implant placement is key to ensuring long-term success. This study compares two methods for determining landmarks for implant placement: using bone-fixed screws (Group 1) versus using remaining teeth that need to be extracted (Group 2).

Study Procedure:

1. Pre-surgery: Patients will undergo general health screenings and a CT scan to plan the surgery.
2. Surgery: Patients will be assigned to:

   1. Group 1: Patients with fewer than 3 remaining teeth or teeth with mobility greater than grade 1, including at least one tooth in the front and one in the back on each side, will have bone screws placed on the bone as landmarks for implant placement using the dynamic navigation system.
   2. Group 2: Patients with at least 3 remaining teeth, with mobility no greater than grade 1, and at least one tooth in the front and one in the back on each side, will use these teeth as landmarks for implant placement.

Post-surgery Evaluation: After surgery, the implant deviation from the planned implant data will be assessed. This will measure the accuracy of the implant placement by comparing the actual position of the implants with the planned position.

Benefits and Risks:

1. Benefits:

   1. Improved accuracy in implant placement using the Dynamic Navigation System.
   2. Cost of using the Dynamic Navigation System and the cost of bone screws for patients without sufficient remaining teeth are covered by the study.
   3. Scientific contribution to improving implant placement methods for future patients.
2. Risks:

   1. Surgical risks including infection, pain, swelling, and potential implant failure, which can occur even without the use of the dynamic navigation system.
   2. Radiation exposure from imaging tests, particularly CBCT scans, will be required. Even if patients do not participate in this study, the CBCT scan is a standard part of the implant placement procedure, and the radiation exposure from CBCT is minimal and within safe limits.
   3. Slight increase in surgery time, typically 2-5 minutes longer than traditional surgery, for preparation and calibration of the navigation system to ensure its proper functionality.
   4. For Group 1 participants, bone screws (4-6 screws) will be placed along the jaw arch where the implants are to be positioned. These screws serve as reference points for the navigation system.

Confidentiality:

All patient information will be kept strictly confidential. Health data and study outcomes will only be used for research purposes and will not be shared with any third parties without the patient's consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are fully edentulous or have partial edentulism and are in need of full arch prosthesis rehabilitation.
* Aged 18 years and older.
* Individuals in good general health (American Society of Anesthesiologists (ASA) class I or II)
* Willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Any serious medical (ASA class III or IV) or psychiatric conditions.
* Pregnant or breastfeeding women.
* General or Local Health Conditions Affecting Surgery: Systemic/local conditions that affect surgical healing, wound healing, and bone integration or use of medications such as steroids, bisphosphonates, or other drugs affecting bone health; smoking more than 10 cigarettes per day; acute infections at the planned implant site that have not been treated.
* Patients with a limited mouth opening of less than 40mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Angular Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the angular Deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Global Platform Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the global platform deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Global Apical Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the global apical deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Platform Depth Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the platform depth deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Apical Depth Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the apical depth deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Platform Bucco-lingual Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the platform bucco-lingual deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Platform Mesiodistal Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the platform mesiodistal deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Apical Bucco-lingual Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the apical bucco-lingual deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Apical Mesiodistal Deviation | The assessment of implant deviation will be measured immediately after surgery
  The primary outcome measure for this study is to evaluate the apical mesiodistal deviation in implant placement when using the dynamic navigation system with bone screw landmarks (Group 1) versus remaining teeth landmarks (Group 2). Implant deviation is defined as the difference between the planned implant positions and the actual placement based on the navigation system. This outcome will help assess the precision of implant placement and compare the two groups for improved accuracy in full arch rehabilitation procedures.
Calibration Time | Calibration time will be recorded during the pre-surgical phase of the implant procedure, immediately before implant placement, in both groups.
  This outcome measure evaluates the calibration time required for the dynamic navigation system before implant placement, comparing Group 1 (bone screw landmarks) and Group 2 (remaining teeth as landmarks). Calibration time is measured from the moment the system is set up to the point where it is ready to guide implant placement. This time frame includes adjustments and validation of the system to ensure accurate implant positioning.
  The primary goal is to compare the calibration times between the two groups to evaluate if the use of bone screws (Group 1) or remaining teeth (Group 2) as landmarks affects the calibration time required by the dynamic navigation system.

CONTACTS AND LOCATIONS:
Overall Officials: Nhiem Cao Tran, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - Dental Center, Ho Chi Minh City
  - Van Hanh General Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
We intend to share IPD regarding the deviation in implant positioning from planned data and the calibration times recorded during the surgical procedures. No personally identifiable information (PII) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date: After study completion End Date: 12 months after study completion
Access Criteria: The IPD and supporting information will be accessible to researchers, regulatory bodies, and other authorized individuals involved in the study. Access will be granted to those who have received approval from the ethics committee or relevant regulatory authorities. These individuals will be able to access the data via a secure, password-protected portal or system provided by the study team. All users will be required to sign a data sharing agreement to ensure confidentiality and compliance with the relevant data protection regulations.